CLINICAL TRIAL: NCT02561520
Title: Safety and Efficacy of Autologous Platelet Rich Plasma and Platelet Poor Plasma Eye Drops in the Treatment of Ocular Graft-Versus-Host Disease
Brief Title: Safety and Efficacy of Autologous PRP and PPP Eye Drops in the Treatment of Ocular GVHD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not enroll participants is being withdrawn from the system.
Sponsor: Ladan Espandar (Other)
Responsible Party: Sponsor-Investigator, Ladan Espandar, Assisant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15070211
Record Dates: First submitted 2015-09-17; First posted 2015-09-28 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Graft-versus-host Disease
Keywords: platelet rich plasma; platelet poor plasma; ocular GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRP and PPP (Experimental): PRP eye drops and PPP eye drops will be prepared from patient's own blood by Magellan technology. Patients will receive eye drops in sterile amber glass droppers. Patients will be instructed to keep refrigerated each bottle after opening for 7 days and keep frozen the unopened bottles up to 30 days.
  Interventions: Biological: PRP eye drops; Biological: PPP eye drops

INTERVENTIONS:
Biological: PRP eye drops — Eye drops 4x a day, patients will start this eye drop first.
  Other Names: Platelet rich plasma
Biological: PPP eye drops — Eye drops 4x a day, patients will start this eye drops after PRP.
  Other Names: Platelet poor plasma

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous Platelet Rich Plasma (PRP) and Platelet Poor Plasma (PPP) eye drops four times a day in the treatment of ocular graft versus host disease (O-GVHD). In addition to their current medication (except autologous serum drops), patients will receive PRP and PPP drops.

DETAILED DESCRIPTION:
Ocular involvement can be quite symptomatic in patients with chronic graft-versus-host disease (GVHD). The impact of ocular GVHD on quality of life (QOL) in patients with chronic GVHD has been studied in a prospective, multicenter, longitudinal, observational study and showed that ocular GVHD affects 57% of patients within 2 years of chronic GVHD diagnosis. Strong evidence suggested that ocular GVHD is associated with worse overall health-related QOL. Significant worsening of vision-related QOL in ocular GVHD has been reported. Ocular GVHD is devastating and there is no effective treatment available so far. The importance of this study is that for the first time in the nation, our institute will evaluate the safety and efficacy of topical autologous blood product (PRP and PPP) to treat ocular surface disease associated with ocular GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with study assessments for the full duration of the study.
* Diagnosis of ocular GVHD.
* Minimum corneal fluorescein staining of 4 (NEI grading scheme, 0-15) in at least one eye.
* In good stable overall health.

Exclusion Criteria:

* Remission from primary cancer in more than 5 years.
* History of thrombocytopenia (platelet<50,000) in the last 2 weeks before study entry.
* Ocular or periocular malignancy.
* Significant change, as judged by the PI, in systemic immunosuppressive regimen before 2 weeks of study entry.
* Any change in dosage of tetracycline compounds (tetracycline, doxycycline, and minocycline) within the last month.
* Any change in frequency of preserved anti-glaucoma medications before 2 weeks of study entry.
* Current use of topical steroids more than twice a day.
* Change in frequency of topical cyclosporine and/or topical kineret within the last month.
* Signs of current infection, including fever and current treatment with antibiotics.
* Intra-ocular surgery or ocular laser surgery within the last 3 months.
* Has worn contact lenses, except for bandage contact lens or rigid gas permeable lens or scleral contact lens, for the last 2 weeks prior to the study or would be unable to stay off contact lenses for the study duration.
* Any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 8 Weeks
  Safety and tolerability of topical autologous PRP and PPP four times a day will be monitored by the occurrence of systemic and ocular adverse events in addition to symptoms directly related to the instillation or use of the autologous blood products. The severity of each adverse event and relation to the study medication will be graded possibly, probably, or definitely related. Tolerability measures will be graded from trace to severe using a direct query method at each visit.

SECONDARY OUTCOMES:
Efficacy of topical autologous PRP and PPP as measured by the National Eye Institute (NEI) grading scale | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing signs of dry eye in ocular GVHD, cornea fluorescein staining will be used using NEI grading system.
Efficacy of topical autologous PRP and PPP as measured by Tear Film Break Up Time (TBUT) | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing signs of dry eye in ocular GVHD,Tear Film Break Up Time (TBUT) will be used.
Efficacy of topical autologous PRP and PPP as measured by Schirmer Test I | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing signs of dry eye in ocular GVHD, Schirmer test without topical anesthetic will be used.
Efficacy of topical autologous PRP and PPP as measured by expression of cellular markers of inflammation using real-time polymerase chain reaction (RT-PCR) | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing signs of dry eye in ocular GVHD, expression of cellular markers of inflammation such as (intercellular adhesion molecule-1 (ICAM-1), interleukin IL-1b, IL-2, IL-6, IL-8, IL-10, IL-17, IL-23, interferon IFN-g and tumor necrosis factor TNF-α) will be used using real-time polymerase chain reaction (RT-PCR) on schirmer filter papers.
Efficacy of topical autologous PRP and PPP as measured by expression of cellular markers of inflammation using flow cytometry (FC) | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing signs of dry eye in ocular GVHD, expression of cellular markers of inflammation such as (intercellular adhesion molecule-1 (ICAM-1), interleukin IL-1b, IL-2, IL-6, IL-8, IL-10, IL-17, IL-23, interferon IFN-g and tumor necrosis factor TNF-α) will be used using flow cytometry (FC) on schirmer filter papers.
Efficacy of topical autologous PRP and PPP as measured by Ocular Surface Disease Index (OSDI) questionnaire | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing symptoms of dry eye in ocular GVHD by Surface Disease Index (OSDI) questionnaire
Efficacy of topical autologous PRP and PPP as measured by National Eye Institute-Visual Function Questionnaire (NEI-VFQ-25) | 8 weeks
  To evaluate the efficacy of topical autologous PRP and PPP four times a day in reducing symptoms of dry eye in ocular GVHD by National Eye Institute-Visual Function Questionnaire (NEI-VFQ-25)

CONTACTS AND LOCATIONS:
Overall Officials: Ladan Espandar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Eye Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided